CLINICAL TRIAL: NCT04228159
Title: The Effectiveness of Perturbation Training With Balance Tutor, Compared to Balance and Strengthening Exercise, on Falls Rate Among Elderly at Risk of Falling
Brief Title: Perturbation Training Compared to Balance and Strengthening Exercise, for Elderly at Risk of Falling
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clalit Health Services (Other)
Collaborators: MediTouch Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: fall prevention BT
Record Dates: First submitted 2020-01-13; First posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2019-12

CONDITIONS: Fall Prevention
Keywords: Accidental Falls, Frail Elderly, Physical Therapy Specialty

STUDY DESIGN:
Intervention Model Description: randomized control trial. Older adults at moderate and high risk of falling will be recruited among Clalit patients referred to one of three physical therapy clinics, or other clinics nearby, neither by physician referral due to gait abnormality or following the physiotherapist diagnosis. Potential participants fulfilling the inclusion criteria and not meeting the exclusion criteria will sign informed consent and continue with baseline assessment. Those not wishing to participate will continue with routine care. Once the baseline assessment is completed, participants will be randomized into one of two intervention groups using computer random allocation software. Participants in both groups will attend physical therapy clinics twice a week for a total of 14 sessions. Each session will last 30 minutes. General information regarding fall prevention will be delivered to all participants using Clalit brochures and electronic prescriptions
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perturbation training (Experimental): Session1 - baseline assessment (detailed above) Session2 - 13 - each session will begin with reassessment and documentation of balance tutor parameters for each participant as were calibrated at the end of previous session.
  After reassessment the training program will include:
  * Warm up - walking without perturbation.
  * Perturbation during standing position.
  * Perturbation during walking.
  * Perturbation during tandem position.
  * Perturbation with vestibular stimulation.
  * Rest according to patient needs The relative duration of each component, as well as intensity and frequency of perturbations, will be adjusted to each individual according to his ability, reassessment parameters and progression.
  Session14 - full reassessment of all baseline examinations including: Mini-BESTest, ABC scale, PASE, and number of falls.
  Interventions: Device: Balance Tutor Biofeedback Rehabilitation System
- Balance and strengthening exercise (Active Comparator): Session1 - baseline assessment (detailed above).
  Session2 - 13 - each session will include:
  * Warm up (free walking or cycling).
  * Static balance exercise - standing position. Exercise will be performed using different bases of support (narrow, tandem, and one leg stance), eyes open/closed, unstable surfaces, functional and cognitive dual task, and vestibular stimulation.
  * Dynamic balance exercise - walking position. Exercise will be performed using different bases of support (narrow, tandem, and one leg stance), eyes open/closed, unstable surfaces, functional and cognitive dual task, and vestibular stimulation.
  * Strengthening exercise - general strengthening, particularly for lower limb.
  * Cool down. Level of difficulty and duration of each component will be adjusted to each individual according to his ability and progression.
  Session14 - full reassessment of all baseline examinations including: Mini-BESTest, ABC scale, PASE, and number of falls.
  Interventions: Other: Balance and strengthening exercise

INTERVENTIONS:
Device: Balance Tutor Biofeedback Rehabilitation System — Balance Tutor system is a unique technology which allows for several postural control ability assessments as well as reactive response training in both standing and walking using controlled perturbation in simple task or multitask performance. Together with proactive training the system allows for optimal rehabilitation outcome and recovery
  Arms: Perturbation training
Other: Balance and strengthening exercise — exercise training programs for fall prevention including walking and balance exercises, functional tasks, strength, flexibility and endurance
  Arms: Balance and strengthening exercise

SUMMARY:
One third of adults over 65 and 50% of adults above 80 years old fall at list once a year. In some cases, falls result in fractures, hospitalization, functional limitations, depression, morbidity and mortality. Strong evidence support exercise training programs for fall prevention, while several studies examined the effect of perturbation training on risk of fall. The aim of this study is to evaluate the effectiveness of a perturbation training program with unexpected perturbation using balance tutor on falls and injuries among elderly at risk of falling, compared to balance and strengthening exercise.

ELIGIBILITY:
Inclusion Criteria:at least one fall during the last 12 months; age 65-85; mini-mental state examination score 24 and above allowing cognitive ability to understand simple instructions ; Time Up and Go (TUG), assessing balance, walking ability and fall risk, scored 13 and above ; ability to read Hebrew or Arabic; and the ability to walk independently 10 meters.

-

Exclusion Criteria:progressive neurological conditions (Parkinson, Multiple sclerosis, CVA); severe orthopedic conditions including lower limb or spine fractures and surgeries in the past 12 months prior to baseline; blindness; Arrhythmia; uncontrolled chronic disease (i.e., hypertension, diabetes, ischemic heart disease); diagnosed severe osteoporosis with a history of fracture during the past 3 years prior to baseline; active cancer during the past three years prior to baseline; lack of availability in the coming two months for completing the treatment protocol

-

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-11-25 (Actual); Primary Completion 2021-05-25 (Estimated); Study Completion 2022-05-25 (Estimated)

PRIMARY OUTCOMES:
rate of falls and fallers | falls and fallers rates during 12-months following end of treatment
hip fractures and hospitalizations rates due to falls | hip fractures and hospitalizations rates due to falls during12-months following end of treatment

SECONDARY OUTCOMES:
Mini-BESTest | end of treatment-last visit in physical therapy clinic
  Balance assessment according to Balance Evaluation Systems Test. The Mini-BESTest is a 14 item test scored on a 3-level ordinal scale. The total score is 28 while a lower score indicates severe balance impairment
Activities-Specific Balance Confidence Scale (ABC scale) | 12 months after end of treatment
  The ABC scale is a 16-item self-report measure in which patients rate their balance confidence for performing activities. Items are rated on a rating scale that ranges from 0-100; 0 represents "no confidence" and 10 represents "complete confidence".
Physical Activity Scale for the Elderly (PASE) | 12 months after end of treatment
  The PASE measures the level of self-reported physical activity in individuals aged 65 years or older and is comprised of items regarding occupational, household, and leisure activities during the previous 7-days period

CONTACTS AND LOCATIONS:
Overall Officials: Shlomit Yaron, MD, Principal Investigator — Clalit Health Services
Locations (3):
- Israel (3):
  - Clalit HealthCare services, Beersheba
  - Clalit Healthcare Services, Holon
  - Clalit HealthCare Services, Nazareth

IPD SHARING:
Plan to Share IPD: No